CLINICAL TRIAL: NCT05655052
Title: The Effect of Virtual Reality Glasses and Distraction Cards on Women's Pain, Anxiety and Satisfaction Level in Intrauterine Device Application'
Brief Title: The Effect of Virtual Reality Glasses Pain, Anxiety and Satisfaction Level in Intrauterine Device Application'
Acronym: Virtual
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mine Gokduman Keles (Other Government)
Responsible Party: Sponsor-Investigator, Mine Gokduman Keles, Midwifery, Turkish Ministry of Health, Kahramanmaras Provincial Health Directorate
Organization: Turkish Ministry of Health, Kahramanmaras Provincial Health Directorate (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TurkishMoHKahramanmaras
Record Dates: First submitted 2022-11-15; First posted 2022-12-16 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Virtual Reality; Pain; Anxiety; Distraction Cards
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: : A randomized controlled trial
Who Masked: Care Provider
Masking Description: According to the AP Polyclinic admission sequence number and from the list determined by randomization (determined from the www.randomizer.org site), which group it is in will be determined. Study and control group assignments will be made.
  It will be applied by the health personnel working in the Family Planning Counseling Polyclinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- working grup 1: Virtual Reality (VR) Group (Experimental): From the preparation stage of the IUD until the IUD application process is completed, after the internet connection is provided with a smart phone for the image, by clicking on the youtube.com link, Relaxation (https://www.youtube.com/watch?v=H1iboKia3AQ) nature video will be provided and virtual reality glasses will be provided.
  Virtual reality glasses to be used in the research are not a medical device. This device is a technological glasses that works with compatible smartphones. The practice of watching nature videos with VR during the IUD application with this device is within the framework of midwifery care practices and is not a treatment option for any treatment method, tool or disease. Although the video watched with VR has no effect on medical treatment and care within the framework of midwifery care, it does not have any harmful effects on women. The participant can withdraw from this study at any time without giving any reason.
  Interventions: Device: Virtual Reality (VR) Group
- Working Group 2: Distraction Cards Implementation Group (Experimental): From the preparation stage of the IUD procedure to the completion of the IUD application process, distraction cards containing five optical illusion figures, one of the distraction techniques, will be shown to the women by the researcher . Distraction cards consist of picture cards with various hidden pictures and patterns. These hidden pictures and patterns are such that individuals can only see when they look carefully. During the process, the women will focus on the cards and be distracted by asking what they see on the cards by communicating face-to-face with the researcher women about the pictures and shapes they see on the cards. Thus, it is thought that the cards with optical figures on the distraction cards will enable women to focus and reduce pain and anxiety. Display of cards will take approximately 3-5 minutes
  Interventions: Device: Group using distraction cards
- Control Group (No Intervention): Unlike the study group, women included in the control group will not only be shown video watching applications with virtual glasses and distraction cards. The maintenance and applications in the routine IUD application will be done exactly.

INTERVENTIONS:
Device: Virtual Reality (VR) Group — At the beginning of the study, the women who applied for the IUD procedure will be interviewed, and then the following procedures will be applied; Informed consent of all women will be obtained about the study.
  * An introductory information form will be filled in for women in all three groups.
  * While the Intervention Group 1 IUD is being applied, a nature video will be watched with Virtual Glasses.
  * Distraction Cards will be shown while the Intervention Group 2 IUD is being administered.
  * The Control Group will be given routine IUD application and care.
  Arms: working grup 1: Virtual Reality (VR) Group
Device: Group using distraction cards — At the beginning of the study, the women who applied for the IUD procedure will be interviewed, and then the following procedures will be applied; Informed consent of all women will be obtained about the study.
  * An introductory information form will be filled in for women in all three groups.
  * While the Intervention Group 1 IUD is being applied, a nature video will be watched with Virtual Glasses.
  * Distraction Cards will be shown while the Intervention Group 2 IUD is being administered.
  * The Control Group will be given routine IUD application and care.
  Arms: Working Group 2: Distraction Cards Implementation Group

SUMMARY:
The aim of this study is to examine the effects of virtual reality glasses and distraction cards, which are cognitive behavioral techniques, on women's pain, anxiety and satisfaction levels. It is aimed to reduce your anxiety level, reduce pain level and increase feelings of satisfaction by showing you a nature video with Virtual Reality Glasses or showing distraction cards so that you can spend this process more comfortably while IUD is being applied. The following questions are expected to be answered in this research: When virtual reality glasses and distraction cards are applied during the IUD procedure; (1) Does it affect the woman's pain level? (2) Does it affect the woman's anxiety level? (3) does it have an effect on women's satisfaction? In addition, it is aimed to reveal the effectiveness of virtual reality glasses and distraction cards in the IUD application process, which is one of the modern family planning methods in midwifery applications, and to bring a non-invasive and cost-effective option into practice.

DETAILED DESCRIPTION:
The proportion of women who want to use Family Planning in the world in the last two decades has reached approximately 1.1 billion and has shown a significant increase . Despite this increasing demand, it is seen that there has been a slow increase of 3.2 in the ratio of family planning (FP) needs met by modern contraceptive methods for women of reproductive age in the last ten years. The reasons for this slow increase include limited access to modern contraceptive methods, women's prejudice about some methods, and low quality of available services . In addition, WHO reported that almost half of pregnancies in developing countries between 2015 and 2019 were unwanted pregnancies , and recommended effective FP counseling and the use of more modern contraceptive methods to prevent this . In Turkey, the Ministry of Health provides individuals with free access to modern FP methods. Despite this, according to 2018 data of the Turkey Demographic and Health Survey (TNSA), it has been reported that 49% use modern methods in the use of FP method, and the Intrauterine Device (IUD) is among the most effective modern methods with a rate of 14% . Among the factors affecting the use of the IUD; women's perception of pain during the application and the fact that it can be applied in certain centers .

In addition, it has been reported in the literature that women perceive pain during IUD application. In these studies, pain; especially used in the stages of IUD application; It is reported that it is detected during tenaculum insertion, measurement with a hysterometer, and finally during IUD insertion. For this reason, there is a need for applications to reduce the pain associated with the IUD application, which is the modern FP method of women. Again, it is assumed that women will experience anxiety before the IUD application as in other medical procedures . It is seen in the literature that there are studies to alleviate the perceived pain in IUD application . In addition, it is expected that the applications made to women for the symptoms such as pain and anxiety related to the applications in the field of health will increase their satisfaction . In this context, there are studies in the literature showing that virtual reality glasses and distraction cards, which are cognitive behavioral techniques, are used during medical procedures, reducing the perception of pain and reducing the level of anxiety. . Although virtual reality glasses are a technological device, they have been widely used in the medical field in hospitals. Virtual reality glasses to be used in the research are not a medical device. This device is a technological glasses that works with compatible smartphones. The applications to be made with this device are within the framework of midwifery care applications and are not a treatment method, mediator or treatment option for any disease and do not have any harmful effects. Again, the cards with optical illusion figures on the distraction cards enable women to focus and reduce pain and anxiety.

No study has been found in the literature examining the effects of virtual reality glasses and distraction techniques on pain, anxiety and satisfaction levels in IUD application. However, in line with the results of the study, it is thought that the IUD procedure will have a positive effect on reducing the perceived pain and anxiety of women and increase satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-45,
* IUD applied,

Exclusion Criteria:

* Having visual and auditory disabilities,
* Use of misoprostol during the procedure,
* Pre-procedure pain medication use,
* Pre-procedure anxiety medication use.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — IUD applied,
Enrollment: 37 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Pulse Rate and Oxygen Saturation | ria application restriction averages 20 minutes
  The pulse rate and saturation values of women will be evaluated physiologically using the sensor compatible planet 50n LT model pulse oximeter (Nellcor COVIDIEN SPO 2) device.
Verbal Category (SKO) | Before the examination; (2) Speculum insertion; (3) Application of the tenaculum to the cervix; (4) During IUD insertion; (5) It will be evaluated five times in total, 15 minutes after the IUD administration (5).
  Verbal Category Scale (SCA) (Appendix 4): The Verbal Category Scale is also called the Simple Descriptive Scale, and this scale is based on the patient's choice of the most appropriate word to describe the pain condition. Pain severity ranges from mild to unbearable. In this scale, he used the words "mild", "disturbing", "severe", "very severe", "unbearable" to describe the severity of pain (Appendix-5). The individual is asked to choose the appropriate category for his situation.
Numerical Pain Rating Scale (SAAS) | Before the examination; (2) Speculum insertion; (3) Application of the tenaculum to the cervix; (4) During IUD insertion; (5) It will be evaluated five times in total, 15 minutes after the IUD administration (5).
  Numerical pain rating scale (SARS) is used to evaluate pain severity. In the numerical evaluation scale, pain ranges from 0 (absence of pain) to 10 (unbearable pain).
State Anxiety Scale (STAI TX-I) | Before and after IUD procedure
  items are answered by marking one of the options such as (1) none, (2) a little, (3) a lot, (4) a lot, depending on the severity of the emotion or behavior. There are two types of expressions in the scale. These are reversed or straight forward expressions. reversed expressions; positive emotions express, while direct expressions express negative emotions. When scoring reverse expressions, those with a weight of 1 are converted to 4, and those with a weight of 4 are converted to 1. In the State Anxiety Scale; There are ten reversed statements, items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20. When scoring, the reversed and direct statements are summed. ints.
Newcastle Nursing Care Satisfaction Scale (NHMS) | ria application restriction averages 20 minutes
  The scale is a 5-point Likert-type scale consisting of 19 items covering nursing care. All items of the Newcastle Nursing Care Satisfaction Scale are positive. In the scoring used to determine the degree of satisfaction, there are statements such as "Not at all Satisfied=1 point, Slightly Satisfied=2 points, Fairly Satisfied=3 points, Very Satisfied=4 points, Extremely Satisfied=5 points". The scores given to the questions of all items marked on the score evaluation scale are added together. The maximum score obtained from the scale is 95, and the minimum score is 19. Evaluation is made by converting the total score obtained from the scale to 100.
Virtual Reality Glasses Application Question | ria application restriction averages 20 minutes
  Virtual Reality Glasses Application Question,It was created by scanning the literature by the researcher.

CONTACTS AND LOCATIONS:
Locations (1):
- TurkishMoHKahramanmarasPH, Kahramanmaraş, Turkey (Türkiye)

REFERENCES:
- [Background] Grimes DA, Lopez LM, Manion C, Schulz KF. Cochrane systematic reviews of IUD trials: lessons learned. Contraception. 2007 Jun;75(6 Suppl):S55-9. doi: 10.1016/j.contraception.2006.12.004. Epub 2007 Feb 16. PMID 17531618
- [Background] Dina B, Peipert LJ, Zhao Q, Peipert JF. Anticipated pain as a predictor of discomfort with intrauterine device placement. Am J Obstet Gynecol. 2018 Feb;218(2):236.e1-236.e9. doi: 10.1016/j.ajog.2017.10.017. Epub 2017 Nov 8. PMID 29079143
- [Background] Gemzell-Danielsson K, Jensen JT, Monteiro I, Peers T, Rodriguez M, Di Spiezio Sardo A, Bahamondes L. Interventions for the prevention of pain associated with the placement of intrauterine contraceptives: An updated review. Acta Obstet Gynecol Scand. 2019 Dec;98(12):1500-1513. doi: 10.1111/aogs.13662. Epub 2019 Jun 27. PMID 31112295
- [Result] Akdemir Y, Karadeniz M. The relationship between pain at IUD insertion and negative perceptions, anxiety and previous mode of delivery. Eur J Contracept Reprod Health Care. 2019 Jun;24(3):240-245. doi: 10.1080/13625187.2019.1610872. Epub 2019 May 16. PMID 31094575
- [Result] Hylton J, Milton S, Sima AP, Karjane NW. Cold Compress for Intrauterine Device Insertional Pain: A Randomized Control Trial. Womens Health Rep (New Rochelle). 2020 Aug 4;1(1):227-231. doi: 10.1089/whr.2020.0056. eCollection 2020. PMID 33786484
- [Derived] Toker E, Gokduman Keles M. The Impact of Virtual Reality with Relaxation Music and Distraction Cards on Pain, Anxiety, and Satisfaction Levels of Women with an Intrauterine Device: A Randomized Controlled Trial. J Midwifery Womens Health. 2025 Nov 14. doi: 10.1111/jmwh.70048. Online ahead of print. PMID 41235692
- See also: Home/Newsroom/Fact sheets/Detail/Family planning/contraception method — https://www.who.int/news-room/fact-sheets/detail/family-planning-contraception
- See also: WHO. New estimates show worldwide fall in unintended pregnancies since 1990-1994. 2020. — https://www.who.int/news/item/23-07-2020-new-estimates-show-worldwide-fall-in-unintended-pregnancies-since-1990-1994
- See also: High rates of unintended pregnancies linked to gaps in family planning services: New WHO study — https://www.who.int/news/item/25-10-2019-high-rates-of-unintended-pregnancies-linked-to-gaps-in-family-planning-services-new-who-study
- See also: TNSA. Türkiye Nüfus ve Sağlık Araştırması 2018 Ne Söylüyor? 2018 — http://www.sck.gov.tr/wp-content/uploads/2020/08/TNSA2018_ana_Rapor.pdf